CLINICAL TRIAL: NCT04000347
Title: A Study of Efficacy of Benzoyl Peroxide Regimens in Treatment of Unpleasant Foot Odor
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to covid 19 outbreaks, the study are suspended.
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: benzoylperoxide_PK
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Benzoyl Peroxide; Foot Dermatoses
Keywords: benzoyl peroxide; Pitted keratolysis; Foot Odor
MeSH Terms: conditions — Foot Dermatoses

STUDY DESIGN:
Who Masked: Participant
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Single blind controlled trial between participants, drug preparing team, doctors, investigators, and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2.5% benzoyl peroxide (Active Comparator): 43 patients with 2.5% benzoyl peroxide gel
  Interventions: Drug: 2.5% benzoyl peroxide gel
- 5% benzoyl peroxide (Active Comparator): 43 patients with 5% benzoyl peroxide gel
  Interventions: Drug: 5% benzoyl peroxide gel

INTERVENTIONS:
Drug: 2.5% benzoyl peroxide gel — 2.5% benzoyl peroxide gel was given to patients for 2 weeks
  Arms: 2.5% benzoyl peroxide
Drug: 5% benzoyl peroxide gel — 5% benzoyl peroxide gel was given to patients for 2 weeks
  Arms: 5% benzoyl peroxide

SUMMARY:
This study aimed to study the efficacy of topical 2.5% benzoyl peroxide, compared to 5% benzoyl peroxide in treatment of unpleasant foot odor, which was considered as major problem related to pitted keratolysis.

DETAILED DESCRIPTION:
Introduction Pitted keratolysis is a common skin disease, caused by various gram-positive bacteria including Corynebacterium species, Kytococcus sedentarius, Dermophilus congolensis and Actinomyces species. These bacteria create small tunnels in the stratum corneum, causing pitted lesions at plantar areas. This condition is frequent accompanied by feet malodor and is commonly found in young male adults, especially in soldiers, miners and athletes. The reported prevalence of pitted keratolysis among naval cadets in Thailand was 38.7%. Predisposing factors related to pitted keratolysis are pedal hyperhidrosis and prolonged feet occlusion. Although this condition is generally not painful, our previous study in 2018 revealed adversely affects patients' quality of life.

Regarding treatment modalities of pitted keratolysis, various medications and life-style modification have been recommended. Previous studies revealed efficacy of topical choices, including benzoyl peroxide gel, clindamycin-benzoyl peroxide gel, glycopyrrolate cream,9 erythromycin gel, clindamycin solution, chlorhexidine scrub4 and mupirocin ointment. Oral antibiotics and botulinum toxin injection were also beneficial in pitted keratolysis. As to life-style modification, wearing cotton socks and opened footwear, and proper hygiene, have also been suggested.

Topical benzoyl peroxide is an over-the-counter drug and is known as off-label medication for pitted keratolysis. It has both aerobic and anaerobic antibacterial properties due to inhibition of various cell functions and the response against bacteria is dose related.15 In addition to antibacterial property, benzoyl peroxide can cause keratolysis. Previous studies by Vlahovic et al. (2009) and Balic et al. (2018) demonstrated efficacy of combination of 1% clindamycin and 5% benzoyl peroxide gel in pitted keratolysis. However, study of efficacy of topical benzoyl peroxide alone or comparison between 2.5% and 5% benzoyl peroxide gel for the treatment of pitted keratolysis is currently limited.

Objective The present study aimed to study the efficacy of topical 2.5% benzoyl peroxide, compared to 5% benzoyl peroxide in treatment of unpleasant foot odor, which was considered as major problem related to pitted keratolysis.

Material and Methods First-year naval rating cadets, who had pedal malodor were invited to enroll in this study. The cadets who previously received any topical treatment including topical antibiotic, antiperspirant or aluminum chloride within 6 months prior to the study were excluded. Consent was informed and obtained from all participants. Participants were assessed for behavioral risk factors and level of foot odor measured by a self-assessed visual analogue scale (VAS), using questionnaires. Clinically examination of feet was done in all subjects by treatment-blinded dermatologists. Subjects were randomly assigned either 2.5% benzoyl peroxide gel or 5% benzoyl peroxide gel for 2 weeks. Benzoyl peroxide gel in this study comprised benzoyl peroxide in a gel base. During the study, using of other topical treatment such as topical antibiotics, antiperspirant or aluminum chloride was not allowed. Participants were advised to apply the drug on their both soles once per day before bedtime to leave it on and were able to regularly participate in physical military training during the study. Two weeks after the treatment, clinical examinations by dermatologists and the cadets' self-assessment questionnaires, including feet odor by using VAS, treatment satisfaction and adverse effects, were used to evaluate the effectiveness. Pitted lesions improvement at plantar areas, evaluated by dermatologists, was divided into no improvement, slight improvement (decrease of pitted lesions at feet for 1 level) and much improvement (decrease of pitted lesions at feet for at least 2 level). Data were analyzed using PASW Statistics version 18 (SPSS, Inc., Chicago, IL, USA). Duration of study: 3 months Study design: Randomized control trial

ELIGIBILITY:
Inclusion Criteria:

* First-year naval rating cadets, who had pedal malodor

Exclusion Criteria:

* The cadets who previously received any topical treatment including topical antibiotic, antiperspirant or aluminum chloride within 6 months prior to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of topical 2.5% benzoyl peroxide, compared to 5% benzoyl peroxide in treatment of unpleasant foot odor | 2 weeks
  Effectiveness was evaluated by the number of patients who had no or minimal foot odor after treatment

SECONDARY OUTCOMES:
Evaluate side effects of topical 2.5% benzoyl peroxide, compared to 5% benzoyl peroxide | 2 weeks
  Side effects was assessed by the percentage of patients developed any side effect such as erythema, burning sensation, pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Almeida HL Jr, Siqueira RN, Meireles Rda S, Rampon G, de Castro LA, Silva RM. Pitted keratolysis. An Bras Dermatol. 2016 Jan-Feb;91(1):106-8. doi: 10.1590/abd1806-4841.20164096. PMID 26982791
- [Result] Makhecha M, Dass S, Singh T, Gandhi R, Yadav T, Rathod D. Pitted keratolysis - a study of various clinical manifestations. Int J Dermatol. 2017 Nov;56(11):1154-1160. doi: 10.1111/ijd.13744. Epub 2017 Sep 18. PMID 28924971
- [Result] van der Snoek EM, Ekkelenkamp MB, Suykerbuyk JC. Pitted keratolysis; physicians' treatment and their perceptions in Dutch army personnel. J Eur Acad Dermatol Venereol. 2013 Sep;27(9):1120-6. doi: 10.1111/j.1468-3083.2012.04674.x. Epub 2012 Aug 7. PMID 22882561
- [Result] Leeyaphan C, Bunyaratavej S, Taychakhoonavudh S, Kulthanachairojana N, Pattanaprichakul P, Chanyachailert P, Ongsri P, Arunkajohnsak S, Limphoka P, Kulthanan K. Cost-effectiveness analysis and safety of erythromycin 4% gel and 4% chlorhexidine scrub for pitted keratolysis treatment. J Dermatolog Treat. 2019 Sep;30(6):627-629. doi: 10.1080/09546634.2018.1543846. Epub 2018 Dec 11. PMID 30415588
- [Result] Vlahovic TC, Dunn SP, Kemp K. The use of a clindamycin 1%-benzoyl peroxide 5% topical gel in the treatment of pitted keratolysis: a novel therapy. Adv Skin Wound Care. 2009 Dec;22(12):564-6. doi: 10.1097/01.ASW.0000363468.18117.fe. No abstract available. PMID 19935134
- [Result] Bunyaratavej S, Leeyaphan C, Chanyachailert P, Pattanaprichakul P, Ongsri P, Kulthanan K. Clinical manifestations, risk factors and quality of life in patients with pitted keratolysis: a cross-sectional study in cadets. Br J Dermatol. 2018 Nov;179(5):1220-1221. doi: 10.1111/bjd.16923. Epub 2018 Sep 14. No abstract available. PMID 29951993
- [Result] Burkhart CG. Pitted keratolysis: a new form of treatment. Arch Dermatol. 1980 Oct;116(10):1104. No abstract available. PMID 7425659
- [Result] Balic A, Bukvic Mokos Z, Marinovic B, Ledic Drvar D. Tatami Mats: A Source of Pitted Keratolysis in a Martial Arts Athlete? Acta Dermatovenerol Croat. 2018 Apr;26(1):68-70. PMID 29782305
- [Result] Kontochristopoulos G, Sidiropoulou P, Tzanetakou V, Markantoni V, Platsidaki E, Agiasofitou E, Rigopoulos D, Gregoriou S. Managing pitted keratolysis: consider topical glycopyrrolate. Clin Exp Dermatol. 2019 Aug;44(6):713-714. doi: 10.1111/ced.13851. Epub 2018 Dec 4. No abstract available. PMID 30515854
- [Result] Pranteda G, Carlesimo M, Pranteda G, Abruzzese C, Grimaldi M, De Micco S, Muscianese M, Bottoni U. Pitted keratolysis, erythromycin, and hyperhidrosis. Dermatol Ther. 2014 Mar-Apr;27(2):101-4. doi: 10.1111/dth.12064. Epub 2013 May 24. PMID 24703267
- [Result] Greywal T, Cohen PR. Pitted keratolysis: successful management with mupirocin 2% ointment monotherapy. Dermatol Online J. 2015 Aug 15;21(8):13030/qt6155v9wk. PMID 26437161
- [Result] Vazquez-Lopez F, Perez-Oliva N. Mupirocine ointment for symptomatic pitted keratolysis. Infection. 1996 Jan-Feb;24(1):55. doi: 10.1007/BF01780656. No abstract available. PMID 8852468
- [Result] Tamura BM, Cuce LC, Souza RL, Levites J. Plantar hyperhidrosis and pitted keratolysis treated with botulinum toxin injection. Dermatol Surg. 2004 Dec;30(12 Pt 2):1510-4. doi: 10.1111/j.1524-4725.2004.30553.x. PMID 15606827
- [Result] Matin T, Patel P, Goodman MB. Benzoyl Peroxide. 2024 Mar 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537220/ PMID 30725905
- [Result] Burkhart CG, Burkhart CN. Antibacterial properties of benzoyl peroxide in aerobic and anaerobic conditions. Int J Dermatol. 2006 Nov;45(11):1373-4. doi: 10.1111/j.1365-4632.2006.02877.x. No abstract available. PMID 17076732